CLINICAL TRIAL: NCT01103895
Title: Ultrasound Dilution Measurement of Cardiac Output Before and After Adult Cardiopulmonary Bypass
Brief Title: Measurement of Cardiac Output Before and After Cardiopulmonary Bypass.
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-HCE101-4A-H; 2R44HL082022-02 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Output
Keywords: cardiac output; cardiopulmonary bypass; ultrasound dilution

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiac output, the amount of blood pumped by the heart in one minute, will be measured in adults undergoing surgery involving cardiopulmonary bypass. Cardiac output will be measured before and after cardiopulmonary bypass using a device that employs ultrasound dilution technology. The ultrasound dilution cardiac output measurements will be validated or compared with cardiac output measurements made using thermodilution, which is the current "gold standard."

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 21 years
* Patients undergoing surgery involving cardiopulmonary bypass
* Patients instrumented with a thermodilution catheter

Exclusion Criteria:

* Patients aged < 21 years
* Patients undergoing surgery "off pump" (not involving cardiopulmonary bypass)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Measurement of cardiac output before and after cardiopulmonary bypass in adult patients.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cardiac output after cardiopulmonary bypass | Less than 10 minutes
  Cardiac output will be measured using an ultrasound dilution technique and compared with cardiac output measured using thermodilution after the completion of surgical procedures involving cardiopulmonary bypass.

SECONDARY OUTCOMES:
Cardiac output before cardiopulmonary bypass | Less than 10 minutes
  Cardiac output will be measured using an ultrasound dilution technique and compared to cardiac output measured using thermodilution. This will serve as a baseline measurement of the patient's cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Krivitski, PhD, DSc, Principal Investigator — Transonic Systems Inc.; Edward P Nast, MD, Principal Investigator — Arnot Ogden Medical Center
Locations (1):
- Arnot Ogden Medical Center, Elmira, New York, United States

IPD SHARING:
Plan to Share IPD: No